CLINICAL TRIAL: NCT03067974
Title: Intranasal Ketamine for Pediatric Procedural Sedation: a Feasibility Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Initial results did not show benefit.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Vivienne Ng, Physician, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1705414419
Record Dates: First submitted 2017-02-11; First posted 2017-03-01 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Failed Moderate Sedation During Procedure; Ketamine Adverse Reaction
Keywords: ketamine; pediatric; procedural sedation
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Children who meet inclusion and exclusion criteria will be approached for participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intranasal ketamine arm (Experimental): 10mg/kg intranasal ketamine administered one time
  Interventions: Drug: Ketamine Hcl 100Mg/Ml Inj

INTERVENTIONS:
Drug: Ketamine Hcl 100Mg/Ml Inj — 10mg/kg of Ketamine Hcl 100Mg/Ml Inj to be administered intranasally for pediatric procedural sedation

SUMMARY:
The purpose of this study is to evaluate the feasibility of intranasal ketamine for adequate sedation of children undergoing minor procedures in the Emergency Department. An intranasal dose of 10mg/kg will be used in patients requiring procedural sedation. The investigators hypothesize that this dose of intranasal ketamine will be able to provide adequate sedation and analgesia for the physician to successfully complete the planned diagnostic or therapeutic intervention (Pediatr Emer Care 2012;28: 767-70). The primary endpoint will be successful sedation, as defined by the ability to complete the planned procedure without rescue medication, which includes re-dosing of the same medication.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2 years to 7 years who present as patients to the Pediatric Emergency Department at Banner University Medical Center Tucson Campus
* Body weight of 20kg or less (actual, estimated, or measured)
* NPO for four hours or more
* Undergoing various procedures, which are deemed by the treating provider to require procedural sedation for the completion of the procedure.

Exclusion Criteria:

* Discretion of parents
* Discretion of provider
* Body weight greater than 20kg (actual, estimated, or measured)
* Starting Aldrete score <9/10
* Known or suspected psychosis
* Known or suspected central nervous system mass, abnormalities, hydrocephalus, or other condition that would suggest elevated pre-anesthetic cerebrospinal fluid pressure
* Significant elevation in blood pressure
* Known hypersensitivity to ketamine
* Non-English or Spanish speaking

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Successful procedural sedation | The patient will be assessed from the start of procedural sedation medication administration until the completion of the procedural sedation, defined as the patient retuning to baseline (alert and oriented x3 with normal behavior).
  Successful procedural sedation, as defined by the ability to complete the planned procedure without rescue medication, which includes re-dosing of the same medication.

CONTACTS AND LOCATIONS:
Overall Officials: Vivienne Ng, MD, MPH, Principal Investigator — University of Arizona
Locations (1):
- Banner Univsersity Medical Center Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No